CLINICAL TRIAL: NCT06547866
Title: Open Label Phase 2 Study Evaluating the Efficacy and Tolerance of a Zanubrutinib and BGB-11417 Combination in Patients Previously Treated for Waldenström Macroglobulinemia. A FILO Study
Brief Title: Study Evaluating the Efficacy and Tolerance of a Zanubrutinib and BGB-11417 Combination in Patients Previously Treated for Waldenström Macroglobulinemia
Acronym: WAZABI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FILOWM4-WAZABI
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zanubrutinb + BGB-11417 (Experimental): cf intervention
  Interventions: Drug: zanubrutinib + BGB-11417

INTERVENTIONS:
Drug: zanubrutinib + BGB-11417 — The investigational medicinal products (IMP) are Zanubrutinib (BGB- 3111) and BGB-11417.Treatment will be administered for a total of twenty 28 day cycles:
  Cycle 1 with zanubrutinib only
  Cycle 2 with zanubrutinib plus BGB-11417 ramp-up cycle 2, day 1 : 10mg cycle 2, day 2 : 20 mg cycle 2, day 3 : 40mg cycle 2, day 4-7 : 80md daily cycle 2, day 8 and beyond : 160 mg daily
  Cycles 3-20 with zanubrutinib plus BGB-11417 full dose

SUMMARY:
This is a French multicenter open label non-randomized Phase II trial evaluating the efficacy and tolerance of a combination of oral zanubrutinib and BGB-11417 in subjects aged 18 years and older with previously treated Waldenström macroglobulinemia (WM) who require therapy according to the consensus panel criteria from the Second International Workshop on Waldenström's macroglobulinemia.

population : Patients with previously treated Waldenstrom macroglobulinemia

The investigational medicinal products (IMP) are Zanubrutinib (BGB- 3111) and BGB-11417.Treatment will be administered for a total of twenty 28 day cycles:

* Cycle 1 with zanubrutinib only
* Cycle 2 with zanubrutinib plus BGB-11417 ramp-up

  * cycle 2, day 1 : 10mg
  * cycle 2, day 2 : 20 mg
  * cycle 2, day 3 : 40mg
  * cycle 2, day 4-7 : 80md daily
  * cycle 2, day 8 and beyond : 160 mg daily
* Cycles 3-20 with zanubrutinib plus BGB-11417 full dose

DETAILED DESCRIPTION:
study design : Open label, multicenter phase 2 trial

population : Patients with previously treated Waldenstrom macroglobulinemia

Primary objective :

To evaluate the efficacy of a combination of zanubrutinib and BGB-11417 given for a limited duration of time in Refractory/Relapsing (R/R) WM by the proportion of subjects achieving either a Complete Response (CR) or Very Good Partial Responses (VGPR).duration of time in Refractory/relapsing (R/R) Waldenstrom macroglobulinemia (WM)

Secondary objectives:

* To further evaluate the efficacy of a combination of zanubrutinib and BGB-11417 given for a limited duration of time in R/R WM
* To determine the incidence and severity of serum M-protein (monoclonal IgM) rebound after planned cessation of the combination of zanubrutinib and BGB-11417-101 in R/R WM
* To evaluate the safety and tolerability of a combination of zanubrutinib and BGB-11417 given for a limited duration of time in R/R WM

Sample size : 102 patients Length of study: Inclusion period: 24 months Treatment duration: 18 months (twenty 28-days cycles) Follow-up period: 3 years

Study treatment :

The investigational medicinal products (IMP) are Zanubrutinib (BGB- 3111) and BGB-11417.Treatment will be administered for a total of twenty 28 day cycles:

* Cycle 1 with zanubrutinib only
* Cycle 2 with zanubrutinib plus BGB-11417 ramp-up
* Cycle 2 with zanubrutinib plus BGB-11417 ramp-up

  *cycle 2, day 1 : 10mg
  * cycle 2, day 2 : 20 mg
  * cycle 2, day 3 : 40mg
  * cycle 2, day 4-7 : 80md daily
  * cycle 2, day 8 and beyond : 160 mg daily
* Cycles 3-20 with zanubrutinib plus BGB-11417 full dose

All patient will receive both drugs.

Study procedures:

Screening period:

Assessments may be done up to 28 days before the treatment start and will include:

Clinical assessments

- Medical history, WM history including prior treatment lines, previous IPSS WM score, histology, known cytogenetics and molecular features including MYD88, CXCR4 and TP53 mutational status

* Concomitant therapies
* Complete physical examination, including weight, height, vital signs, ECOG performance status, B symptoms, detailed evaluation of lymph nodes, liver and spleen and infection monitoring (including COVID-19 nasal test)
* IPSS WM score

Biological assessments

* Standard hematology tests including CBC (hemoglobin, WBC count, absolute differential count, platelet count)
* Blood coagulation tests including: prothrombin time, activated cephalin time, fibrinogen, von Willebrand factor (vWF; including vWF antigen [vWF:Ag] and vWF:Activity [WF:Act]; evaluation according to ABO blood group) and FVIII* *If acquired Willebrand syndrome according to hemorrhagic risk assessment, further analysis is encouraged.
* Blood chemistry tests including sodium, potassium, chloride, bicarbonate, fasting glucose, phosphate, blood urea nitrogen (BUN), creatinine, calcium, phosphate, magnesium, total, direct and indirect bilirubin, total protein, albumin, alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT), lactate dehydrogenase (LDH), alkaline phosphatase (PAL), uric acid, C-reactive protein (CRP), beta2microglobulin and pregnancy test
* Troponin; NT-proBNP will be performed on blood
* Serum "M-protein" (monoclonal IgM) quantification based on protein electrophoresis or alternate methods (according to appendix 3), immunofixation, nephelometry, free light chains kappa and lambda, cryoglobulinemia
* IgG, IgA and IgM levels
* Serologies for HBV, HCV and HIV

Cardiovascular assessments:

* Cardiovascular evaluation by investigator:

  o 12-lead ECG and QTc calculation

  o blood pressure after 5 minutes rest, average of 3 measurements separated by ≥ 1 minute.
* Cardiovascular evaluation by cardiologist*:

  * 12-lead ECG with QTc calculation
  * echocardiography
  * 24h Holter ECG monitoring
  * 24h Ambulatory blood pressure monitoring (ABPM)

Imaging assessments:

-Whole-Body CT scan (neck, thorax, abdomen, pelvis) with tumor measurements

Specific assessments:

* BM biopsy* (local laboratory).

  *This can be omitted if already done within the past 3 months.
* BM aspirate for oLocal laboratory for Cytogenetic analysis and FISH for 17p oFILOthèque central laboratory, storage for future analysis: unsorted and CD19+ sorted cells for mutational profile.
* Blood MRD assessment on plasmatic cell-free tumor DNA (FILOthèque central laboratory).

Treatment period

Clinical assessment:

* Concomitant therapies and adverse events, severe adverse events and adverse events of special interest (AE, SAE and AESI)
* Complete physical examination, including evaluation of lymph nodes, liver and spleen

Cardiovascular assessments:

-Cardiovascular evaluation by investigator after 1, 3, 6, 9, 12, 15 and 18 cycles: o12-lead ECG and QTc calculation* oblood pressure after a 5 minute rest, average of 3 measurements separated by ≥ 1 minute.

* The 12-lead ECG by investigator is not mandatory if already done or planned during the cardiology consultation within one month (at cycle 3, 6, 12, and 18)

  -Cardiovascular evaluation by cardiologist after 3, 6, 12, and 18 cycles: ocardiology consultation o24h Holter ECG monitoring* o24h ABPM** oEchocardiography***
* 24h Holter ECG will be repeated only at cycles 3, 6 and 18 (only risk patient)

  * 24h ABMP will be repeated only at cycles 3, 12 and 18

    * Echocardiography will be repeated at cycle 18.

Biological assessments (at day 1 +/- 7 days of each cycle):

* Standard hematology tests including CBC (hemoglobin, WBC count, absolute differential count, platelet count)
* Blood chemistry: including sodium, potassium, chloride, bicarbonate, fasting glucose, phosphate, BUN, creatinine, calcium, phosphate, magnesium, total, direct and indirect bilirubin, total protein, albumin, ALAT, ASAT, LDH, PAL, uric acid, CRP and pregnancy test.

During ramp up period: serum creatinine, sodium, potassium, chloride, bicarbonate, calcemia, phosphoremia, LDH is mandatory before initiation of any ramp up dose of BGB-11417, and 8 and 24 hours after drug intake.

* Troponin and NT-proBNP at cycles 1, 3, 6, 9, 12, 15 and 18
* Serum "M-protein" (monoclonal IgM) quantification based on protein electrophoresis or alternate methods (according to appendix 3) with additional immunofixation (to confirm CR)
* IgG, IgA and IgM levels

Imaging assessments:

-Whole-body CT scan (neck, thorax, abdomen, pelvis) every 24 weeks (6 cycles) i.e. after cycles 3, 6, 12 and 18 in all subjects who had measurable nodal/extranodal disease at screening.

Specific assessments:

-FILOthèque central laboratory: Blood on specific tube for MRD assessment on plasmatic cell-free tumor DNA (at cycles 3, 6, 12 and 18), storage.

Response evaluation:

Throughout the treatment period, especially before "end of treatment (EOT) + 3 months (EVAL 2 ) evaluation":

* if a CR is suspected (negative IF), an unscheduled CT scan should be done followed by biological evaluations including BM biopsy (local laboratory) to confirm CR
* If a VGPR is suspected (≥90% reduction in serum M-protein (monoclonal IgM) level from baseline (but still detectable) and decreased lymphadenopathy/ splenomegaly (if present at baseline), an unscheduled CT scan should be done to confirm VGPR.

Evaluation 1 (EVAL 1): 1 month after the end of treatment This evaluation takes place 1 month after EOT either after completion of cycle 20 or after the last cycle in case of early discontinuation. This evaluation may detect M-protein rebound with or without other features of early progression.

Clinical assessments:

* Concomitant therapies
* AE, SAE and AESI
* Complete physical examination including evaluation of lymph nodes, liver and spleen

Cardiovascular assessments:

-Cardiovascular evaluation by investigator: o12-lead ECG and QTc calculation oBlood pressure after a 5 minute rest, average of 3 measurements separated by ≥ 1 minute

Biological assessments:

* Standard hematology tests including CBC (hemoglobin, WBC count, absolute differential count, platelet count)
* Blood chemistry: sodium, potassium, chloride, bicarbonate, fasting glucose, phosphate, BUN, creatinine, calcium, phosphate, magnesium, total, direct and indirect bilirubin, total protein, albumin, ALAT, ASAT, LDH, PAL, uric acid, CRP, and pregnancy test.
* Serum "M-protein" (monoclonal IgM) quantification based on protein electrophoresis or alternate methods (according to appendix 3) with additional immunofixation (to confirm a CR)
* IgG, IgA and IgM levels

Evaluation 2 (=EVAL 2): 3 months after the end of treatment This evaluation takes place 3 months after EOT either after completion of cycle 20 or after the last cycle in case of early discontinuation. This evaluation may detect M-protein rebound with or without other features of early progression.

Clinical assessments:

* Concomitant therapies
* AE, SAE and AESI
* Complete physical examination, including evaluation of lymph nodes, liver and spleen

Cardiovascular assessments:

-Cardiovascular evaluation by investigator: o12-lead ECG and QTc calculation oBlood pressure after 5 minutes rest, average of 3 measurements separated by ≥ 1 minute

-Cardiovascular evaluation by a cardiologist: oCardiology consultation o24h Ambulatory blood pressure monitoring (ABPM) oEchocardiography

Biological assessments:

* Standard hematology tests including CBC (hemoglobin, WBC count, absolute differential count, platelet count)
* Blood chemistry: sodium, potassium, chloride, bicarbonate, fasting glucose, phosphate, BUN, creatinine, calcium, phosphate, magnesium, total, direct and indirect bilirubin, total protein, albumin, ALAT, ASAT, LDH, PAL, uric acid, CRP
* NT-proBNP
* Serum "M-protein" (monoclonal IgM) quantification based on protein electrophoresis or alternate methods (according to appendix 3) with additional immunofixation (to confirm a CR)
* IgG, IgA and IgM levels

Imaging and BM assessments:

* Whole body CT scan
* BM biopsy (local laboratory) if not performed during the treatment period for CR or progression.
* BM aspirate (FILOthèque central laboratory) for storage and analysis for molecular studies without CD19 sorting.
* Blood collected on specific tube (FILOthèque central laboratory) for assessment of plasmatic cell-free tumor DNA

Evaluation in case of suspected CR At any time throughout the study, especially before "EOT evaluation" when a CR is suspected based on a negative immunofixation, an additional evaluation should be realized in order to confirm the CR.

This additional evaluation includes primarily:

* Repeated screening for cryoglobulinemia, in patients known to have significant cryoglobulinemia at screening.
* CT scan

Then, if both immunofixation and CT scan are consistent with CR, a biological assessment should be scheduled with:

-BM biopsy (local laboratory)

Evaluation in case of suspected VGPR At any time throughout the study, especially before "EOT evaluation", when a VGPR is suspected based on ≥90% reduction in M-protein (monoclonal IgM) level from baseline (but still detectable) and decreased lymphadenopathy/splenomegaly (if present at baseline), an additional evaluation should be realized in order to confirm the VGPR.

This additional evaluation includes:

* Repeated screening for cryoglobulinemia, in patients known to have significant cryoglobulinemia at screening.
* CT scan: to confirm the reduction of deep-seated lymphadenopathy and splenomegaly (if present at baseline)

Evaluation in case of progression during treatment and follow-up period

* BM biopsy optional (local laboratory)
* BM aspirate, indicated according to study only in case of progression for :
* local laboratory: cytogenetics and FISH for 17p
* FILOthèque central laboratory: storage of unsorted and CD19+ sorted cells for molecular analyzes.
* Blood collected on specific tube for assessment of plasmatic cell-free tumor DNA (FILOthèque central laboratory).

Post-treatment follow-up period after EVAL 2 Two follow-up evaluations scheduled at 1 month (EVAL 1) and at 3 months (EVAL 2) have been already detailed above. Thereafter, all patients enrolled in the study will be followed until progression or death every 3 months the first year (FU6, FU9 and FU12), then every 6 months for a total follow up period of three years (FU18, FU24, FU30 and FU36).

Clinical assessments:

* Concomitant therapies
* AE, SAE and AESI
* Complete physical examination, evaluation of lymph nodes, liver and spleen.

Cardiovascular assessments:

* Cardiovascular evaluation by investigator o12-lead ECG and QTc calculation oblood pressure after 5 minutes rest, average of 3 measurements separated by ≥ 1 minute
* Cardiovascular evaluation by a cardiologist (only at FU36) ocardiology consultation o24h ABPM oEchocardiography

Biological assessments:

* Standard hematology tests including CBC (hemoglobin, WBC count, absolute differential count, platelet count).
* Blood chemistry: sodium, potassium, chloride, bicarbonate, fasting glucose, phosphate, BUN, creatinine, calcium, phosphate, magnesium, total, direct and indirect bilirubin, total protein, albumin, ALAT, ASAT, LDH, PAL, uric acid, CRP
* NT-proBNP (only FU36)
* Serum "M-protein" (monoclonal IgM) quantification based on protein electrophoresis or alternate methods (according to appendix 3) with additional immunofixation (to confirm a CR)
* IgG, IgA and IgM levels

Imaging and BM assessments:

* Whole body CT scan if clinically indicated, especially in case of progression.
* BM biopsy (local laboratory)
* BM aspirate, indicated according to study, only in case of progression

Premature end of treatment (PEOT) A visit will be performed 4 weeks (EVAL 1) and 3 months (EVAL 2) after the last treatment day for patients who discontinue treatment prematurely and for patients withdrawing their consent (if possible),

In case of PEOT for disease progression, patients will be evaluated

End of study (EOS) The end of study becomes effective after the end of the last study visit of the last patient enrolled once the FU36 visit has been achieved. The end of study visit corresponds to the last follow-up visit (FU36). For patients withdrawing consent during the follow up period, no end of study visit is required.

Observational study For all patients if they consent, the survival data will be collected every year for an observational study, in the e-CRF (Survival date and/or event date) until death, for OS analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥ 18-year-old.
2. Have received at least 1 prior line of treatment (excluding treatment with any BTKi or Bcl-2 antagonist, see non-inclusion criteria).
3. Provide written informed consent.
4. Have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3.
5. Have adequate renal function defined as creatinine clearance ≥ 50 mL/min as determined by the Cockroft-Gault equation.
6. Have adequate hepatic function defined as:

   * total serum bilirubin ≤ 1.5 × ULN, unless bilirubin rise is due to Gilbert's syndrome or non-hepatic cause.
   * alanine aminotransferase (ALAT) < 2 × ULN
   * aspartate aminotransferase (ASAT) < 2 × ULN,
7. Have adequate BM function defined as:

   * absolute neutrophil count ≥ 1x109/L
   * platelet count ≥ 75 x109/L
8. For women of childbearing potential, a negative pregnancy test must be documented prior to enrollment.

   * A woman is considered of childbearing potential, ie, fertile, following menarche and until becoming postmenopausal unless permanently sterile. Permanent sterilization methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.
   * A post-menopausal state is defined as no menses for 12 months without an alternative medical cause.
9. Agree to use a highly effective form of contraception with sexual partners throughout study participation (for female and male patients who are fertile). Patients using hormonal contraceptives (eg, birth control pills or devices) must use a barrier method of contraception (eg, condoms) as well.
10. Ability to comply with study procedures, in the Investigator's opinion.
11. Patient covered by any social security system

Exclusion Criteria:

1. Have previously been treated with a BTK inhibitor.
2. Have been previously treated with a bcl-2 antagonist.
3. Have active central nervous system (CNS) disease as evidenced by cytology or pathology. In the absence of clinical signs of CNS disease, a lumbar puncture is not mandatory.
4. Have significant or active cardiovascular disease:

   * stage III to IV congestive heart failure (CHF) as determined by the New York Heart Association (NYHA) classification system for heart failure and/or with left ventricular ejection fraction < 50%
   * myocardial infarction within 6 months before study treatment.
   * unstable angina within 6 months before study treatment.
   * uncontrolled atrial arrhythmia.
   * history of clinically significant ventricular arrhythmias (e.g sustained ventricular tachycardia, ventricular fibrillation, torsades de pointe).
   * uncontrolled hypertension.
   * history of stroke or intracranial hemorrhage within 180 days before the first dose of study drugs
   * QTcF interval > 450 ms on screening electrocardiogram (ECG) evaluation.
5. Have a history of stroke or intracranial hemorrhage within 6 months before first dose of study drug, have a history of a severe bleeding disorder such as hemophilia A, hemophilia B, von Willebrand disease, or history of spontaneous bleeding requiring blood transfusion or other medical intervention:

   * patients with constitutional hemophilia or von Willebrand's disease will be excluded.
   * patients with acquired hemophilia will be excluded.
   * Requires ongoing treatment with warfarin or warfarin derivatives.
   * patients with acquired von Willebrand's disease related to WM can be included. i) if bleeding manifestations are considered as non-clinically significant (i.e.grade 2 or below) ii) or if bleeding manifestations have been corrected by plasma exchange
6. Have received live vaccine within 4 weeks of inclusion.
7. Receive other concomitant investigational therapy.
8. Have a history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, or hepatic condition that, in the opinion of the Investigator, would adversely affect a subject's participation in the study.
9. Have currently active, clinically significant Child-Pugh Class B or C hepatic impairment.
10. Present an inability or difficulty swallowing capsules/tablets, malabsorption syndrome, or any disease or medical condition significantly affecting gastrointestinal function.
11. Have a known allergy to either xanthine oxidase inhibitors or rasburicase or zanubrutinib (patients at risk for G6PD deficiency may be screened before enrolment).
12. Are pregnant or lactating. Women of childbearing potential must agree to use highly effective contraception from the time of signing informed consent until end-of-treatment visit,

    ≥90 days after last dose of BGB-11417-101 and Zanubrutinib. Male patients must be abstinent, vasectomized, or agree to the use of barrier contraception in combination with other methods.
13. Have a history of other active malignancies requiring treatment within 3 years of study entry, with exception of (1) localized basal cell or squamous cell carcinoma of the skin, (2), adequately treated in situ endometrial carcinoma, (3) incidental histology finding of prostate carcinoma, (4) previous malignancy confined and treated locally (surgery or other modality) with curative intent.
14. Be known to be positive for HIV.
15. Present evidence of other clinically significant uncontrolled condition(s) including, but not limited to:

    * uncontrolled and/or active systemic infection (viral, bacterial or fungal) including COVID-19
    * chronic hepatitis B virus (HBV) or hepatitis C (HCV) requiring treatment. Note: subjects with serologic evidence of prior vaccination to HBV (i.e. hepatitis B surface [HBs] antigen negative-, anti-HBs antibody positive and anti-hepatitis B core [c] antibody negative) or positive anti-HBc antibody from intravenous immunoglobulins (IVIG) may participate. Patients with serologic evidence of prior resolved infection can be included according to recommendations .
16. Suffer from any condition or illness that, in the opinion of the Investigator or medical monitor, would compromise patient safety or interfere with the evaluation of the safety of the study drugs.
17. Have received or consumed any of the following within 3 days prior to the first dose of study drugs:

    * grapefruit or grapefruit products.
    * Seville oranges (including marmalade containing Seville oranges).
    * star fruit.
18. Have received a treatment with any of the following prior to the first dose of study drugs:

    * ≤7 days steroid therapy with anti-neoplastic intent.
    * ≤ 7 days or 5 half-lives (whichever is longer) of any moderate or strong CYP3A4 inhibitor and ≤ 14 days or 5 half-lives, (whichever is longer) of moderate or strong CYP3A4 inducer before the first dose of study drugs.
    * allogeneic or autologous stem cell transplantation or CAR-T cell therapy less than 3 months before the first dose of study drugs.
19. Severe or debilitating pulmonary disease.
20. Major surgery within 4 weeks of the first dose of study drug.
21. Active and/or ongoing autoimmune anemia and/or autoimmune thrombocytopenia (eg, idiopathic thrombocytopenia purpura).
22. Ongoing alcohol or drug addiction or any psychiatric condition(s) which would compromise ability to comply with study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | twenty 28-days cycles
  Number of subjects achieving a CR or VGPR at any time during the course of treatment

SECONDARY OUTCOMES:
Overall response rate (ORR) | at any time during the course of study treatment (twenty 28-days cycles)
  Number of subjects achieving a best response (CR, VGPR, PR or minor response)
Major response rate (MRR) | at any time during the course of study treatment (twenty 28-days cycles)
  Number of subjects achieving a best response (CR, VGPR or PR)
Time to response (TTR) | From start to end of treatment (twenty 28-days cycles)
  time to achieve of at least a minor response
Progression free survival (PFS) | From start of treatment to end fo Fup (twenty 28-days cycles + 3 years Fup)
  time to disease progression or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Kamel Laribi, MD, Principal Investigator — CH Le Mans
Locations (37):
- France (37):
  - AMIENS - CH Amiens Picardie Site Sud, Amiens
  - Angers Chu, Angers
  - ANNECY - CH Annecy Genevois, Annecy
  - ARGENTEUIL - Centre hospitalier Victor Dupouy, Argenteuil
  - BAYONNE - CH de la Côte Basque - Hématologie, Bayonne
  - BESANCON - Hôpital Jean Minjoz, Besançon
  - Bordeaux-Institut Bergonié, Bordeaux
  - CAEN - CHU Caen - IHBN, Caen
  - Clermont-Ferrand - Chu Estaing, Clermont-Ferrand
  - CRETEIL - CHU Henri Mondor, Créteil
  - DIJON - Hôpital François Mitterrand, Dijon
  - Grenoble - CHUGA - Hématologie Clinique, Grenoble
  - La Roche Sur Yon - Chd Vendee, La Roche-sur-Yon
  - Le Mans CH, Le Mans
  - LILLE GHICL - Hôpital Saint Vincent de Paul, Lille
  - LILLE CHU - Hôpital Claude Huriez, Lille
  - LYON-Centre Léon Bérard, Lyon
  - MARSEILLE - Institut Paoli-Calmettes, Marseille
  - MONTPELLIER - Hôpital Saint-Eloi - Hématologie Clinique, Montpellier
  - Mulhouse - Ghrmsa, Mulhouse
  - NANTES - Hôpital Hôtel Dieu - Hématologie Clinique, Nantes
  - ORLEANS - CHR - Hématologie, Orléans
  - APHP - Hôpital Pitié Salpêtrière - Hématologie, Paris
  - PERPIGNAN - CH St Jean - Hématologie Clinique, Perpignan
  - Bordeaux Pessac, Pessac
  - LYON HCL - CH Lyon Sud, Pierre-Bénite
  - POITIERS - Hématologie et Thérapie Cellulaire, Poitiers
  - Reims Chu, Reims
  - RENNES - CHU Pontchaillou - Hématologie Clinique, Rennes
  - ROUEN - Centre Henri Becquerel - Service Hématologie Clinique, Rouen
  - Strasbourg - Icans, Strasbourg
  - Toulouse - IUCT Oncopole - Service d'Hématologie, Toulouse
  - TOURS - Hôpital Bretonneau, Tours
  - NANCY - CHU Brabois, Vandœuvre-lès-Nancy
  - Vannes - Chba, Vannes
  - VERSAILLES - Hôpital André Mignot, Versailles
  - Villejuif Igr, Villejuif

IPD SHARING:
Plan to Share IPD: No